CLINICAL TRIAL: NCT01146418
Title: Follow-up Protocol to Collect the Outcome and Safety of Frozen-thawed Embryo Transfer (FTET) Cycles After Cryopreservation of Embryos in Clinical Study P06029 (Phase 3; Protocol No. P06031)
Brief Title: Frozen-thawed Embryo Transfer (FTET) Cycle Follow-up Protocol (P06031)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P06031
Record Dates: First submitted 2010-06-11; First posted 2010-06-17 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Infertility
Keywords: Reproductive Techniques, Assisted; Follicle Stimulating Hormone, Human; Fertilization In Vitro
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corifollitropin alfa 150 μg (Experimental): Participants in Base Study P06029 received a single injection of 150 ug corifollitropin alfa on Stimulation Day 1 and daily injections of placebo-recFSH from Stimulation Days 1 through 7. No medication or investigational product was administered in Follow-Up Study P06031.
  Interventions: Biological: Corifollitropin alfa
- recFSH 300 IU (Active Comparator): Participants in the reference group in Base Study P06029 received a single injection of placebo for corifollitropin alfa on Stimulation Day 1 and daily injections of 300 IU recFSH on Stimulation Days 1 through 7. No medication or investigational product was administered in Follow-Up Study P06031.
  Interventions: Biological: recFSH (follitropin beta)

INTERVENTIONS:
Biological: Corifollitropin alfa — Single injection of 150 μg corifollitropin alfa administered under protocol P06029
  Arms: Corifollitropin alfa 150 μg
Biological: recFSH (follitropin beta) — Daily recFSH 300 IU administered under protocol P06029.
  Other Names: Follistim® AQ Cartridge
  Arms: recFSH 300 IU

SUMMARY:
The purpose of this follow-up study is to collect the outcome and safety of FTET cycles after the embryos are cryopreserved in P06029 (NCT01144416). P06029 was a study in which a single injection of corifollitropin alfa (SCH 900962) was compared with daily recombinant follicle stimulating hormone (recFSH) injections in women aged 35 to 42 years undergoing controlled ovarian stimulation (COS) prior to in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have provided written informed consent for the trial.
* Participant must have cryopreserved embryo(s) in trial P06029 (NCT01144416) of which at least one embryo is thawed for use in a subsequent FTET cycle.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 307 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2013-07-24 (Actual); Study Completion 2014-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boostanfar R, Gates D, Guan Y, Gordon K, McCrary Sisk C, Stegmann BJ. Efficacy and safety of frozen-thawed embryo transfer in women aged 35 to 42 years from the PURSUE randomized clinical trial. Fertil Steril. 2016 Aug;106(2):300-305.e5. doi: 10.1016/j.fertnstert.2016.03.041. Epub 2016 Apr 16. PMID 27090863

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period 1 consists of participants from Base Study P06029 (NCT01144416) randomized to treatment groups corifollitropin alfa or recombinant follicle stimulating hormone (recFSH). Period 2 consists of participants from base study enrolled in Follow-Up Study P06031. Period 3 consists of infants born to expectant mothers in Follow-Up Study P06031.
Groups:
- Corifollitropin Alfa 150 μg Women/Expectant Mothers: Participants in Base Study P06029 (NCT01144416) received a single injection of 150 ug corifollitropin alfa on Stimulation Day 1 and daily injections of placebo-recFSH from Stimulation Days 1 through 7. Eligible participants from the base study could enroll in Follow-Up Study P06031. No medication or investigational product was administered in this follow-up study.
- recFSH 300 IU Women/Expectant Mothers: Participants in the reference group in Base Study P06029 (NCT01144416) received a single injection of placebo for corifollitropin alfa on Stimulation Day 1 and daily injections of 300 IU recFSH on Stimulation Days 1 through 7. Eligible participants from the base study could enroll in Follow-Up Study P06031. No medication or investigational product was administered in this follow-up study.
- Corifollitropin Alfa 150 μg Live-Born Infants: Infants born to eligible participants who received a single injection of 150 μg corifollitropin alfa in Base Study P06029 (NCT01144416) were followed for safety and efficacy in Follow-Up Study P06031 according to standard practice.
- recFSH 300 IU Live-Born Infants: Infants born to eligible participants who received daily 300 IU recFSH in Base Study P06029 (NCT01144416) were followed for safety and efficacy in Follow-Up Study P06031 according to standard practice.
Period: Base Study P06029 (NCT01144416)
Arm/Group | Corifollitropin Alfa 150 μg Women/Expectant Mothers | recFSH 300 IU Women/Expectant Mothers | Corifollitropin Alfa 150 μg Live-Born Infants | recFSH 300 IU Live-Born Infants
Started | 694 | 696 | 0 | 0
Completed | 632 (Participants who underwent ET in base study) | 647 (Participants who underwent ET in base study) | 0 | 0
Not Completed | 62 | 49 | 0 | 0
Period: Women/Expectant Mother Follow Up
Arm/Group | Corifollitropin Alfa 150 μg Women/Expectant Mothers | recFSH 300 IU Women/Expectant Mothers | Corifollitropin Alfa 150 μg Live-Born Infants | recFSH 300 IU Live-Born Infants
Started | 157 (Participants from Base Study P06029 with at least one embryo thawed for use in FTET cycle.) | 150 (Participants from base study P06029 with at least one embryo thawed for use in FTET cycle.) | 0 | 0
Participants With Embryo Transfer (ET) | 151 | 147 | 0 | 0
Participants With an Ongoing Pregnancy | 52 (Ongoing pregnancy defined as intra-uterine pregnancy with fetal heart beat on USS 10 weeks after ET) | 50 (Ongoing pregnancy defined as intra-uterine pregnancy with fetal heart beat on USS 10 weeks after ET) | 0 | 0
Completed | 113 (Participants with ET transfer who completed follow-up study) | 110 (Participants with ET transfer who completed follow-up study) | 0 | 0
Not Completed | 44 | 40 | 0 | 0
Period: Live-Born Infant Follow Up
Arm/Group | Corifollitropin Alfa 150 μg Women/Expectant Mothers | recFSH 300 IU Women/Expectant Mothers | Corifollitropin Alfa 150 μg Live-Born Infants | recFSH 300 IU Live-Born Infants
Started | 0 | 0 | 61 | 56
Completed | 0 | 0 | 55 (Infants who completed follow up) | 51 (Infants who completed follow up)
Not Completed | 0 | 0 | 6 | 5

BASELINE CHARACTERISTICS:
Population: All Subjects Evaluable, restricted to subjects with ET
Groups:
- Total: Total of all reporting groups
Arm/Group | Corifollitropin Alfa 150 μg Women/Expectant Mothers | recFSH 300 IU Women/Expectant Mothers | Total
Number analyzed (Participants) | 151 | 147 | 298
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (2.1) | 38.3 (2.2) | 38.4 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 147 | 298
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥1 Vital Pregnancy (Cumulative Vital Pregnancy Rate)
Description: The cumulative vital pregnancy rate was defined as the number of participants with at least 1 vital pregnancy in a controlled ovarian stimulation (COS) cycle in Base Study P06029 or a frozen-thawed embryo transfer (FTET) in Follow Up Study P06031, divided by the total number of participants in each Full Analysis Set (FAS) treatment group. A vital pregnancy was defined as an intrauterine pregnancy with fetal heart tones assessed at least 35 days (≥5 weeks) after embryo transfer (ET).
Time Frame: Assessed at least 35 days after ET in COS cycle in Base Study P06029 or an FTET cycle in Follow-Up Study P06031 (up to 2 years)
Population: Full Analysis Set (FAS) population consisted of all randomized participants who received corifollitropin alfa or recFSH in Base Study P06029.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Corifollitropin Alfa 150 μg Women/Expectant Mothers | recFSH 300 IU Women/Expectant Mothers
Number analyzed (Participants) | 694 | 696
Percentage of Participants | 31.1 [27.7 to 34.7] | 33.0 [29.6 to 36.7]
Statistical Analysis 1: Comparison: Corifollitropin Alfa 150 μg Women/Expectant Mothers vs recFSH 300 IU Women/Expectant Mothers; Test type: Superiority or Other; Clopper-Pearson method; Difference calculated using generalized linear model including covariates for treatment group and age class as stratified (≤38 yrs vs >38 yrs); Estimated Difference = -1.8, 95% CI 2-sided [-6.5 to 3.0]

2. Secondary Outcome: Percentage of Participants With ≥1 Live Birth (Cumulative Live-Birth Rate)
Description: The cumulative live-birth rate was defined as the number of participants with at least 1 live birth after ET in a COS cycle in Base Study P06029 or an FTET in Follow-Up Study P06031, divided by the total number of participants in each FAS treatment group.
Time Frame: From approximately 10 weeks after ET in Base Study P06029 or FTET in Follow-Up Study P06031 up to time of delivery (up to 2 years)
Population: FAS population consisted of all randomized participants who received corifollitropin alfa or recFSH in Base Study P06029.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Corifollitropin Alfa 150 μg Women/Expectant Mothers | recFSH 300 IU Women/Expectant Mothers
Number analyzed (Participants) | 694 | 696
Percentage of Participants | 28.2 [24.9 to 31.8] | 29.5 [26.1 to 33.0]
Statistical Analysis 1: Comparison: Corifollitropin Alfa 150 μg Women/Expectant Mothers vs recFSH 300 IU Women/Expectant Mothers; Test type: Superiority or Other; Clopper-Pearson method; [statistical method as in outcome 1, analysis 1]; Estimated difference = -1.2, 95% CI 2-sided [-5.7 to 3.4]

ADVERSE EVENTS:
Time Frame: From approximately 10 weeks after ET in Base Study P06029 or FTET in Follow-Up Study P06031 up to 12 weeks after birth in current follow-up study (up to 2 years)
Groups:
- Corifollitropin Alfa 150 μg Participants With ET; Corifollitropin Alfa 150 μg Expectant Mothers: Participants in Base Study P06029 (NCT01144416) received a single injection of 150 ug corifollitropin alfa on Stimulation Day 1 and daily injections of placebo-recFSH from Stimulation Days 1 through 7. Eligible participants from the base study could enroll in Follow-Up Study P06031. No medication or investigational product was administered in this follow-up study.
- recFSH 300 IU Participants With ET; recFSH 300 IU Expectant Mothers: Participants in the reference group in Base Study P06029 (NCT01144416) received a single injection of placebo for corifollitropin alfa on Stimulation Day 1 and daily injections of 300 IU recFSH on Stimulation Days 1 through 7. Eligible participants from the base study could enroll in Follow-Up Study P06031. No medication or investigational product was administered in this follow-up study.
- Corifollitropin Alfa 150 μg Follow-up Fetuses/Infants: Infants born to eligible participants who received a single injection of 150 μg corifollitropin alfa in Base Study P06029 (NCT01144416) were followed for safety and efficacy in Follow-Up Study P06031 according to standard practice.
- recFSH 300 IU Follow-up Fetuses/Infants: Infants born to eligible participants who received daily 300 IU recFSH in Base Study P06029 (NCT01144416) were followed for safety and efficacy in Follow-Up Study P06031 according to standard practice
Arm/Group | Corifollitropin Alfa 150 μg Participants With ET | recFSH 300 IU Participants With ET | Corifollitropin Alfa 150 μg Expectant Mothers | recFSH 300 IU Expectant Mothers | Corifollitropin Alfa 150 μg Follow-up Fetuses/Infants | recFSH 300 IU Follow-up Fetuses/Infants
Serious Adverse Events (participants affected / at risk) | 4/151 | 3/147 | 34/52 | 29/50 | 15/61 | 17/56
Other Adverse Events (participants affected / at risk) | 64/151 | 45/147 | 26/52 | 19/50 | 18/61 | 21/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 150 μg Participants With ET (N=151) | recFSH 300 IU Participants With ET (N=147) | Corifollitropin Alfa 150 μg Expectant Mothers (N=52) | recFSH 300 IU Expectant Mothers (N=50) | Corifollitropin Alfa 150 μg Follow-up Fetuses/Infants (N=61) | recFSH 300 IU Follow-up Fetuses/Infants (N=56)
Tachycardia foetal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Single umbilical artery (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal heart rate abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Complication of delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pregnancy with advanced maternal age (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Previous caesarean section (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Caesarean section (Surgical and medical procedures) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Myomectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Congenital lacrimal passage anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital ovarian anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bradycardia foetal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amniotic cavity infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Funisitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital pyelocaliectasis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactoid syndrome of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Selective abortion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 150 μg Participants With ET (N=151) | recFSH 300 IU Participants With ET (N=147) | Corifollitropin Alfa 150 μg Expectant Mothers (N=52) | recFSH 300 IU Expectant Mothers (N=50) | Corifollitropin Alfa 150 μg Follow-up Fetuses/Infants (N=61) | recFSH 300 IU Follow-up Fetuses/Infants (N=56)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (5) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (11) | 5 (6) | 2 (3) | 6 (6) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 10 (10)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 14 (17) | 11 (15) | 1 (2) | 3 (5) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 3 (3)
Vomiting neonatal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (4)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Afterbirth pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Labour pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 37 (38) | 22 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 13 (18) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.